CLINICAL TRIAL: NCT06169254
Title: High-frequency Transcranial Random Noise Stimulation (Hf-tRNS) for Sleep Disturbances in Neurocognitive Disorders Due to Vascular Disease
Brief Title: High-frequency tRNS for Sleep Disturbances in Neurocognitive Disorders Due to Vascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.074
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sleep Disorders, Circadian Rhythm; Cognitive Impairment; Vascular Dementia
Keywords: Aging; Transcranial current stimulation; Sleep disturbance; Randomized clinical trial
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Cognitive Dysfunction; Dementia, Vascular; Parasomnias | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-frequency Transcranial Random Noise Stimulation (Hf-tRNS) (Active Comparator): The stimulation parameters of hf-tACS include: 20 minutes at 101-640 Hz, 2 milliamps.
  Interventions: Device: Transcranial current stimulation (tCS)
- Transcranial alternating current stimulation (tACS) (Active Comparator): The stimulation parameters of HD-tACS include: 20 minutes at 40 Hz, 2 milliamps.
  Interventions: Device: Transcranial current stimulation (tCS)
- Sham transcranial current stimulation (tCS) (Sham Comparator): In sham condition, the stimulation only last for 30 seconds with the electrodes left in place for a further 20 minutes.
  Interventions: Device: Transcranial current stimulation (tCS)

INTERVENTIONS:
Device: Transcranial current stimulation (tCS) — Transcranial current stimulation (tCS) is delivered by a battery driven direct current stimulator (DC-Stimulator Plus, NeuroConn, Ilmenau, Germany) through a central anodal electrode surrounded by four return cathodal electrodes.

SUMMARY:
The investigators aim to 1) investigate and compare the safety, efficacy and sustainability of hf-tRNS, tACS and sham transcranial current stimulation (tCS) over left inferior parietal lobe (IPL) in mild neurocognitive disorder due to vascular disease (NCD-vascular) patients with sleep disturbances; 2) examine the relationship between the changes in sleep quality, cognitive function and brain morphometry.

Methods: Chinese right-handed mild NCD-AD patients with sleep disturbances (aged from 60 to 90 years) will be randomly assigned to a 2-week intervention of either hf-tRNS, tACS, or sham tCS, with 10 participants per arm. Before intervention, structural magnetic resonance imaging (MRI) data is used to construct individual realistic head model. Comprehensive assessments, including sleep quality, cognitive performance and blood pressure will be conducted at baseline, 2th week, 6th week and 12th week. Program adherence and adverse effects will be monitored throughout intervention.

DETAILED DESCRIPTION:
This study aims to investigate the feasibility, safety and efficacy of hf-tRNS and tACS over left IPL for sleep disturbances and cognitive dysfunction in mild NCD-vascular patients. It wills also test the program adherence, tolerability and adverse effects of this innovative neurotechonology. Information will be helpful for in-depth understanding the relationship of "sleep disturbances-cognition" and guiding the further studies of sleep medicine and neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, right-handed, aged from 60 to 80 years.
* With at least one cerebrovascular risk factor, e.g., a history of hypertension defined as systolic blood pressure (BP) 140 mm Hg or higher, diastolic BP of 90 mm Hg or higher; or receiving antihypertensive medication.
* Score of Montreal Cognitive Assessment Hong Kong version (HK MoCA) range from 22 to 26 (Lu et al., 2019).
* With preserved functional abilities reflected by a Functional Assessment Questionnaire score of 7 or lower (Hajjar et al., 2020).
* With a medial temporal lobe atrophy (MTA) score < 2
* No interference with independence in everyday activities.

Exclusion Criteria:

* Previous diagnosis of dementia or stroke;
* Past history of bipolar disorders or psychosis;
* Physically frail affecting attendance to training sessions;
* Already attending regular training, such as cognitive behavioral therapy;
* Taking a psychotropic or other medication known to affect cognition (e.g. anti-dementia medication);
* Significant communicative impairments.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | 12 weeks
  The PSQI is a 19-item questionnaire that includes seven areas of subjective sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction (Buysse et al., 1988). Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.77 to 0.83), sensitivity (89.6%), specificity (86.5%)(Buysse et al., 1988). Greater score of PSQI indicates worse sleep quality.
Attentional function | 12 weeks
  Complex attention is measured by attention network test (ANT). The ANT paradigm is run by E-Prime 3.0 software. Within ANT paradigm, there are four types of cue: no cue, center cue, double cue, and spatial cue; and three types of flanker: neutral, congruent, and incongruent. The reaction time (RT) under different types of flanker indicates the efficacy of attention. Greater score indicates lower efficacy of attentional components.
Executive function | 12 weeks
  Executive function is measured by the category verbal fluency test (CVFT). On each trial, the participants will be asked to overtly generate words in the animal category, fruit category and vegetable category as many as possible within 60 seconds. The total number of correct words is used to measure executive function.

SECONDARY OUTCOMES:
Objective assessment of circadian rhythm | 12 weeks
  Actigraphic records were used to quantify sleep-wake cycle and estimate the objective sleep efficiency.
Global cognition | 12 weeks
  Montreal Cognitive Assessment Hong Kong version (HK MoCA), which is validated global assessment sensitive to detect early cognitive dysfunction in neurocognitive disorder. A total score of HK MoCA less than 26 indicates mild cognitive impairment.
Learning and memory function | 12 weeks
  Word-list learning test (WLLT), consisting of ten semantically non-associated words that is presented consecutively over three free trials of immediate recall, a 20-min delayed recall (to prevent recency effects).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna LU, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong Y, Li J, Yuen YS, Yang NS, Li Z, Tang WK, Lu H. Daily high-frequency transcranial random noise stimulation (hf-tRNS) for sleep disturbances and cognitive dysfunction in patients with mild vascular cognitive impairments: A study protocol for a pilot randomized controlled trial. PLoS One. 2024 Oct 23;19(10):e0309233. doi: 10.1371/journal.pone.0309233. eCollection 2024. PMID 39441802